CLINICAL TRIAL: NCT00593190
Title: Intracameral Gas SF6 (Sulfur Hexafluoride) Injection for Acute Hydrops in Keratoconus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Dr. Boris Safianik, Ha'Emek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0097-07-EMC
Record Dates: First submitted 2008-01-01; First posted 2008-01-14 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Hydrops in Keratoconus
MeSH Terms: interventions — Sulfur Hexafluoride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Gas SF6 (Sulfur Hexafluoride)

INTERVENTIONS:
Drug: Gas SF6 (Sulfur Hexafluoride) — ONCE

SUMMARY:
Intracameral Gas SF6 (Sulfur Hexafluoride) Injection for Acute Hydrops in Keratoconus

ELIGIBILITY:
Inclusion Criteria:

* Hydrops

Exclusion Criteria:

* Age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Hydrops resulotion | weeks

CONTACTS AND LOCATIONS:
Locations (1):
- HaEmek Medical Center, Afula, Israel